CLINICAL TRIAL: NCT03467919
Title: The Effect of Micro Fragmented Adipose Tissue (MFAT) on Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Eugene Roh, Director, Sports Ultrasound Medicine, Orthobiologics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 41688
Record Dates: First submitted 2017-12-20; First posted 2018-03-16 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis, Knee; Knee Pain
Keywords: osteoarthritis; stem cell; knee pain; adipose derived stem cell; injection; MFAT; Micro Fragmented Adipose Tissue
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Micro Fragmented Adipose Tissue (MFAT) on Knee Osteoarthritis
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MFAT(Micro Fragmented Adipose Tissue) (Experimental): Intra-articular knee injection of autologous Micro Fragmented Adipose Tissue harvested from the thigh using tumescent lipoaspiration and processing with minimal manipulation. This harvested tissue will then be injected into the patient's knee.
  Micro Fragmented Adipose Tissue: Harvesting of Micro Fragmented Adipose Tissue with intra-articular injection
  Interventions: Biological: Micro Fragmented Adipose Tissue
- Conventional therapy (Active Comparator): Intra-articular injection of corticosteroid (Triamcinolone 40mg).
  Corticosteroid injection: Sham harvesting of adipose tissue without intra-articular injection. Intra-articular injection of corticosteroid.
  Interventions: Biological: Corticosteroid injection

INTERVENTIONS:
Biological: Micro Fragmented Adipose Tissue — Harvesting of Micro Fragmented Adipose Tissue with intra-articular injection
  Other Names: MFAT
  Arms: MFAT(Micro Fragmented Adipose Tissue)
Biological: Corticosteroid injection — Sham harvesting of adipose tissue without intra-articular injection. Intra-articular injection of corticosteroid.
  Arms: Conventional therapy

SUMMARY:
This is a non-surgical trial comparing the clinical and functional outcomes of patients with osteoarthritis treated with Intra-articular injection of Micro Fragmented Adipose Tissue versus conventional therapy of intra-articular injection of corticosteroid.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial to compare outcomes between intra-articular injection of Micro Fragmented Adipose Tissue and intra-articular injection of corticosteroid in patients with mild to moderate osteoarthritis of the knee. Micro Fragmented Adipose Tissue will be harvested at the subcutaneous tissue by lipoaspiration. Once fat tissue is obtained, it will be processed with minimal manipulation in the clinic room.

To be considered for participation in this study, patients must have radiographic evidence of mild to moderate osteoarthritis of medial and/or lateral weight-bearing compartments (Kellgren-Lawrence Grade 2 or 3). In addition, patients must meet several inclusion/exclusion criteria to be randomized and included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35 and 75 years-old
* Diagnosis of pre-existing osteoarthritis of the joint by Kellgren-Lawrence Grade 2 or 3.
* Working understanding of the English language and able to fully understand the procedure
* Capable of providing informed consent
* Able to complete online, in-person or phone surveys for the purposes of follow-up
* Capable of understanding pre- and post-procedure care instructions
* Ambulatory at baseline
* Previous trial and failure of conservative therapy consisting of a minimum of 6 weeks of physical therapy and trial of anti-inflammatory medications if not contraindicated, with or without concomitant bracing and/or injections.

Exclusion Criteria:

* Age < 35 or > 75 years old
* Radiographs demonstrating either no, little or severe osteoarthritis (Kellgren-Lawrence Grade 0, 1 )
* Prior total or partial joint replacement surgery or a surgery involving cartilage regeneration (microfracture, ACI, etc)
* Previous cortisone and/or Hyaluronic acid intra-articular injection within the last 3 months
* Co-morbidity with rheumatologic condition, inflammatory arthritis
* Currently undergoing immunomodulatory therapy
* Uncontrolled endocrine disorder
* BMI >35
* Current diagnosis of osteomyelitis, human immunodeficiency virus (HIV-1, -2) and/or hepatitis C (HCV), infection and poorly controlled diabetes (HgA1C >7.0)
* Pregnancy or planned pregnancy
* previous stem cell injection into treatment joint
* Patient scheduled to undergo any concomitant surgical procedures.
* Coagulopathy or anticoagulant treatment
* Chronic pain involving multiple body parts or opioid medication management

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Y Roh, MD, Principal Investigator — Stanford University; Jason Dragoo, MD, Principal Investigator — Stanford University; Seth Sherman, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 40 participants signed informed consent, 39 received randomized study injection and provided baseline information
Groups:
- MFAT(Micro Fragmented Adipose Tissue): Intra-articular knee injection of autologous Micro Fragmented Adipose Tissue harvested from the thigh using tumescent lipoaspiration and processing with minimal manipulation.
- Conventional Therapy: Intra-articular injection of corticosteroid (Triamcinolone 40mg).
Period: Overall Study
Arm/Group | MFAT(Micro Fragmented Adipose Tissue) | Conventional Therapy
Started | 30 | 10
Received injection | 30 | 10
Started study procedures | 29 | 10
Completed | 27 | 8
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Population: Participants who started study procedures
Groups:
- Total: Total of all reporting groups
Arm/Group | MFAT(Micro Fragmented Adipose Tissue) | Conventional Therapy | Total
Number analyzed (Participants) | 29 | 10 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (11.0) | 57.9 (11) | 57.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 3 | 19
  Male | 13 | 7 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 20 | 7 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 10 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change in Knee Injury and Osteoarthritis Outcomes Score (KOOS) Score - Pain
Description: Patient reported outcome measure that reports a normalized score (100 indicating no symptoms and 0 indicating extreme symptoms).
Time Frame: Baseline, 3, 6, 12, and 24 months
Population: Participants with data at the respective time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Participants: Combined analysis of all participants.
Arm/Group | MFAT(Micro Fragmented Adipose Tissue) | Conventional Therapy | All Participants
Number analyzed (Participants) | 29 | 10 | 39
score on a scale
  Baseline | 64.4 (17.0) | 62.5 (21.3) | 63.9 (17.9)
  Change at 3 Months: number analyzed (Participants) | 27 | 9 | 36
  Change at 3 Months | 13.2 (16.4) | 8.6 (22.8) | 12.0 (18.0)
  Change at 6 Months: number analyzed (Participants) | 28 | 10 | 38
  Change at 6 Months | 11.1 (13.8) | 6.1 (21.2) | 9.8 (15.9)
  Change at 12 Months: number analyzed (Participants) | 28 | 9 | 37
  Change at 12 Months | 10.8 (23.0) | 14.2 (21.6) | 11.6 (22.4)
  Change at 24 Months: number analyzed (Participants) | 25 | 8 | 33
  Change at 24 Months | 9.6 (18.7) | 14.9 (26.8) | 10.9 (20.6)
Statistical Analysis 1: Comparison: MFAT(Micro Fragmented Adipose Tissue) vs Conventional Therapy; Between-group analysis of change at 3 months; Test type: Other; p = 0.594, two-sample t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: MFAT(Micro Fragmented Adipose Tissue) vs Conventional Therapy; Between-group analysis of change at 6 months; Test type: Other; p = 0.501, two-sample t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 3: Comparison: MFAT(Micro Fragmented Adipose Tissue) vs Conventional Therapy; Between-group analysis of change at 12 months; Test type: Other; p = 0.694, two-sample t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 4: Comparison: MFAT(Micro Fragmented Adipose Tissue) vs Conventional Therapy; Between-group analysis of change at 24 months; Test type: Other; p = 0.611, two-sample t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 5: Comparison: All Participants; Analysis of change at month 3; Test type: Other; p < 0.001, paired t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 6: Comparison: All Participants; Analysis of change at month 6; Test type: Other; p < 0.001, paired t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 7: Comparison: All Participants; Analysis of change at 12 months; Test type: Other; p = 0.003, paired t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 8: Comparison: All Participants; Analysis of change at 24 months; Test type: Other; p = 0.005, paired t-test — The a priori threshold for statistical significance was < 0.05

2. Primary Outcome: Change in Knee Injury and Osteoarthritis Outcomes Score (KOOS) Score - Symptoms
Description: as for outcome 1
Time Frame: Baseline, 3, 6, 12, and 24 months
Population: Participants with data at the respective time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MFAT(Micro Fragmented Adipose Tissue) | Conventional Therapy | All Participants
Number analyzed (Participants) | 29 | 10 | 39
score on a scale
  Baseline | 49.0 (14.3) | 47.5 (19.3) | 48.6 (15.5)
  Change at 3 Months: number analyzed (Participants) | 27 | 9 | 36
  Change at 3 Months | 4.5 (13.3) | 2.8 (24.9) | 4.1 (16.6)
  Change at 6 Months: number analyzed (Participants) | 28 | 10 | 38
  Change at 6 Months | 7.2 (14.7) | 6.1 (16.1) | 7.0 (14.9)
  Change at 12 Months: number analyzed (Participants) | 28 | 9 | 37
  Change at 12 Months | 8.5 (18.1) | 6.7 (17.2) | 8.1 (17.6)
  Change at 24 Months: number analyzed (Participants) | 25 | 8 | 33
  Change at 24 Months | 5.9 (12.2) | 13.8 (16.7) | 7.8 (13.6)
Statistical Analysis 1: Comparison: MFAT(Micro Fragmented Adipose Tissue) vs Conventional Therapy; Between-group analysis of change at 3 months; Test type: Other; p = 0.847, two-sample t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: MFAT(Micro Fragmented Adipose Tissue) vs Conventional Therapy; Between-group analysis of change at 6 months; Test type: Other; p = 0.839, two-sample t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 3: Comparison: MFAT(Micro Fragmented Adipose Tissue) vs Conventional Therapy; Between-group analysis of change at 12 months; Test type: Other; p = 0.791, two-sample t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 4: Comparison: MFAT(Micro Fragmented Adipose Tissue) vs Conventional Therapy; Between-group analysis of change at 24 months; Test type: Other; p = 0.241, two-sample t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 5: Comparison: All Participants; Analysis of change at month 3; Test type: Other; p = 0.149, paired t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 6: Comparison: All Participants; Analysis of change at 6 months; Test type: Other; p = 0.006, paired t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 7: Comparison: All Participants; Analysis of change at 12 months; Test type: Other; p = 0.008, paired t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 8: Comparison: All Participants; Analysis of change at 24 months; Test type: Other; p = 0.002, paired t-test — The a priori threshold for statistical significance was < 0.05

3. Secondary Outcome: Lysholm Score
Description: Patient reported activity outcome measure on a scale of 0-100 (100 is best activity score)
Time Frame: Baseline, 3, 6, 12, and 24 months
Population: Participants with data at the respective time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MFAT(Micro Fragmented Adipose Tissue) | Conventional Therapy | All Participants
Number analyzed (Participants) | 29 | 10 | 39
score on a scale
  Baseline | 60.1 (20.3) | 63.3 (22.2) | 60.9 (20.5)
  Change at 3 Months: number analyzed (Participants) | 27 | 9 | 36
  Change at 3 Months | 10.1 (17.5) | 6.3 (20.6) | 9.1 (18.1)
  Change at 6 Months: number analyzed (Participants) | 28 | 10 | 38
  Change at 6 Months | 12 (16.9) | 3.1 (16.2) | 9.7 (17)
  Change at 12 Months: number analyzed (Participants) | 28 | 9 | 37
  Change at 12 Months | 14 (20.4) | 5.4 (24.2) | 11.9 (21.4)
  Change at 24 Months: number analyzed (Participants) | 25 | 8 | 33
  Change at 24 Months | 10.2 (19.4) | 10.1 (35.4) | 10.2 (23.6)
Statistical Analysis 1: Comparison: MFAT(Micro Fragmented Adipose Tissue) vs Conventional Therapy; Between-group analysis of change at 3 months; Test type: Other; p = 0.633, two-sample t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: MFAT(Micro Fragmented Adipose Tissue) vs Conventional Therapy; Between-group analysis of change at 6 months; Test type: Other; p = 0.158, two-sample t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 3: Comparison: MFAT(Micro Fragmented Adipose Tissue) vs Conventional Therapy; Between-group analysis of change at 12 months; Test type: Other; p = 0.358, two-sample t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 4: Comparison: MFAT(Micro Fragmented Adipose Tissue) vs Conventional Therapy; Between-group analysis of change at 24 months; Test type: Other; p = 0.996, two-sample t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 5: Comparison: All Participants; Analysis of change at 3 months; Test type: Other; p = 0.004, paired t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 6: Comparison: All Participants; Analysis of change at 6 months; Test type: Other; p = 0.001, paired t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 7: Comparison: All Participants; Analysis of change at 12 months; Test type: Other; p = 0.002, paired t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 8: Comparison: All Participants; Analysis of change at 24 months; Test type: Other; p = 0.019, paired t-test — The a priori threshold for statistical significance was < 0.05

4. Secondary Outcome: Veterans RAND 12 (VR-12) Score - Physical
Description: Patient reported quality of life outcome measure. VR-12 scores are reported as T-scores, which are standardized to have a mean of 50 and a standard deviation of 10 in the US population. Higher scores indicate better physical outcomes. Because this is a normalized range, there is theoretically no strict upper or lower bound. Most people will fall somewhere between 20-70 (+/- 3 SD).
Time Frame: Baseline, 3, 6, 12, and 24 months
Population: Participants with data at the respective time point.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | MFAT(Micro Fragmented Adipose Tissue) | Conventional Therapy | All Participants
Number analyzed (Participants) | 29 | 10 | 39
T-score
  Baseline | 42.9 (7.4) | 42.5 (7.0) | 42.8 (7.2)
  Change at 3 Months: number analyzed (Participants) | 27 | 9 | 36
  Change at 3 Months | 3.4 (7.7) | 4.6 (5.0) | 3.7 (7.1)
  Change at 6 Months: number analyzed (Participants) | 28 | 10 | 38
  Change at 6 Months | 4.0 (7.9) | 3.4 (6.2) | 3.8 (7.4)
  Change at 12 Months: number analyzed (Participants) | 28 | 10 | 38
  Change at 12 Months | 5.4 (8.5) | 5 (6.6) | 5.3 (8)
  Change at 24 Months: number analyzed (Participants) | 25 | 8 | 33
  Change at 24 Months | 4.9 (7.8) | 1.8 (9.9) | 4.1 (8.3)
Statistical Analysis 1: Comparison: MFAT(Micro Fragmented Adipose Tissue) vs Conventional Therapy; Between-group analysis of change at 3 months; Test type: Other; p = 0.593, two-sample t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: MFAT(Micro Fragmented Adipose Tissue) vs Conventional Therapy; Between-group analysis of change at 6 months; Test type: Other; p = 0.820, two-sample t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 3: Comparison: MFAT(Micro Fragmented Adipose Tissue) vs Conventional Therapy; Between-group analysis of change at 12 months; Test type: Other; p = 0.867, two-sample t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 4: Comparison: MFAT(Micro Fragmented Adipose Tissue) vs Conventional Therapy; Between-group analysis of change at 24 months; Test type: Other; p = 0.439, two-sample t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 5: Comparison: All Participants; Analysis of change at month 3; Test type: Other; p = 0.004, paired t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 6: Comparison: All Participants; Analysis of change at month 6; Test type: Other; p = 0.003, paired t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 7: Comparison: All Participants; Analysis of change at month 12; Test type: Other; p < 0.001, paired t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 8: Comparison: All Participants; Analysis of change at month 24; Test type: Other; p = 0.008, paired t-test — The a priori threshold for statistical significance was < 0.05

5. Secondary Outcome: Veterans RAND 12 (VR-12) Score - Mental
Description: Patient reported quality of life outcome measure. VR-12 scores are reported as T-scores, which are standardized to have a mean of 50 and a standard deviation of 10 in the US population. Higher scores indicate better mental outcomes. Because this is a normalized range, there is theoretically no strict upper or lower bound. Most people will fall somewhere between 20-70 (+/- 3 SD).
Time Frame: Baseline, 3, 6, 12, and 24 months
Population: Participants with data at the respective time point.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | MFAT(Micro Fragmented Adipose Tissue) | Conventional Therapy | All Participants
Number analyzed (Participants) | 29 | 10 | 39
T-score
  Baseline | 55.9 (8.8) | 58.7 (9.4) | 56.6 (8.9)
  Change at 3 Months: number analyzed (Participants) | 27 | 9 | 36
  Change at 3 Months | -1.6 (8) | -4.3 (10.2) | -2.3 (8.5)
  Change at 6 Months: number analyzed (Participants) | 28 | 10 | 38
  Change at 6 Months | -2.3 (6.4) | -3.5 (8.7) | -2.6 (7)
  Change at 12 Months: number analyzed (Participants) | 28 | 10 | 38
  Change at 12 Months | -2.2 (7.7) | -5.7 (7.5) | -3.1 (7.7)
  Change at 24 Months: number analyzed (Participants) | 25 | 8 | 33
  Change at 24 Months | -0.9 (6) | -2.0 (8.7) | -1.4 (6.6)
Statistical Analysis 1: Comparison: MFAT(Micro Fragmented Adipose Tissue) vs Conventional Therapy; Between-group analysis of change at 3 months; Test type: Other; p = 0.480, two-sample t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: MFAT(Micro Fragmented Adipose Tissue) vs Conventional Therapy; Between-group analysis of change at 6 months; Test type: Other; p = 0.686, two-sample t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 3: Comparison: MFAT(Micro Fragmented Adipose Tissue) vs Conventional Therapy; Between-group analysis of change at 12 months; Test type: Other; p = 0.229, two-sample t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 4: Comparison: MFAT(Micro Fragmented Adipose Tissue) vs Conventional Therapy; Between-group analysis of change at 24 months; Test type: Other; p = 0.564, two-sample t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 5: Comparison: All Participants; Analysis of change at month 3; Test type: Other; p = 0.122, paired t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 6: Comparison: All Participants; Analysis of change at month 6; Test type: Other; p = 0.027, paired t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 7: Comparison: All Participants; Analysis of change at month 12; Test type: Other; p = 0.018, paired t-test — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 8: Comparison: All Participants; Analysis of change at month 24; Test type: Other; p = 0.232, paired t-test — The a priori threshold for statistical significance was < 0.05

6. Other Pre Specified Outcome: MRI Cartilage Scan
Description: Cartilage thickness on MRI using T2-weighted cartilage mapping
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | MFAT(Micro Fragmented Adipose Tissue) | Conventional Therapy
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/10
Other Adverse Events (participants affected / at risk) | 0/30 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT03467919/Prot_000.pdf
  • Statistical Analysis Plan (2025-10-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT03467919/SAP_001.pdf